CLINICAL TRIAL: NCT03165175
Title: Mobile Application for Prescription Drug-Abuse Education (MAPDE)
Acronym: MAPDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Naval Health Research Center (U.S. Federal Agency)
Collaborators: Intelligent Automation, Inc. (Industry)
Responsible Party: Principal Investigator, Suzanne Hurtado, Research Psychologist, GS-13, Naval Health Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HHSN271201500071C
Record Dates: First submitted 2017-05-19; First posted 2017-05-24 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Prescription Drug Abuse (Not Dependent)
Keywords: prescription drug abuse; prescription drug misuse; risk reduction; education; military; mobile application; substance misuse; substance abuse
MeSH Terms: conditions — Substance-Related Disorders; Prescription Drug Misuse; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App + treatment as usual (Experimental): The experimental group will be provided with the prescription drug-abuse education smartphone application in addition to treatment as usual. This educational mobile phone app focuses on helping military members reduce their risk for prescription drug misuse.
  Interventions: Behavioral: prescription drug-abuse education smartphone application
- Treatment as usual (No Intervention): The control group will be provided with treatment as usual, and will also receive a list of resources for help with prescription drug and other substance abuse issues.

INTERVENTIONS:
Behavioral: prescription drug-abuse education smartphone application — As a patient-centered prevention effort, this brief intervention in a mobile phone app format focuses on helping military members reduce their risk for prescription drug misuse. It contains modules to: (1) assess risk for misuse and related behavioral health concerns; (2) provide individualized feedback on risk level; (3) store information on current medications and look up drug interaction and related information; (4) enhance communication and decision-making skills within healthcare and other interpersonal contexts by providing interactive scenarios; (5) teach about the risks of prescription drug misuse; and (6) provide available resources for help with prescription drug misuse.
  Arms: App + treatment as usual

SUMMARY:
The aims of this pilot study are: (1) to assess the feasibility and acceptability of a mobile application to educate military members about the risks of prescription drug misuse; (2) to determine if there is evidence that the mobile application plus treatment as usual reduces the risk of prescription drug misuse and shows differences in related measures compared to treatment as usual among military medical clinic patients currently taking prescription medication; and (3) if evidence of reduced risk is found, to estimate effect sizes for a future effectiveness trial. The pilot study will use a randomized controlled design with two groups. The control group will be provided with treatment as usual (TAU), and the experimental group will be provided with the prescription drug-abuse educational smartphone application in addition to treatment as usual (app + TAU). Self-reported measures of risk of misuse and related attitudes and knowledge will be administered to all participants at baseline, 1 month, and 3 months. The mobile app is a brief intervention designed to help military members to assess their risk for medication misuse and provide individualized feedback on risk level with recommendations for reducing risk. The app also contains other features, including sections in which to store information on current medications and look up drug interactions and provides resources for help.

DETAILED DESCRIPTION:
Subjects:

Eighty active duty participants will be initially recruited for this study. With attrition, the final sample size is expected to be 60. Potential participants will be patients of the pain clinic, deployment health clinic or other clinics, or pharmacy patrons of the Naval Medical Center San Diego (NMCSD) who have currently been prescribed a medication(s) with the potential for misuse. The participants will likely reflect the demographics of the overall Navy population. The sample is also expected to include a variety of racial groups and ranks. A list of prescription medications with the potential for misuse will be used for the medication criterion. The list was developed based on information from the National Institute on Drug Abuse, Commonly Abused Drugs Charts-prescription drugs; the Drug Enforcement Agency; and consultations with Navy pain clinic physicians and a Navy pharmacist.

Methods and Informed Consent Plan:

Study design. The study consists of a randomized controlled design with two groups. The control group will be provided with treatment as usual, and the experimental group will be provided with the prescription drug-abuse education smartphone application in addition to treatment as usual. Repeated measures will be administered to all participants at baseline, 1 month, and 3 months. This study does not propose any modification of, change to or interference with the physician's treatment plan, and the app is not considered a medical device under section 201(h) of the Federal Food, Drug, and Cosmetic Act (FD&C Act). Study results will also be used to determine estimates of intervention effect sizes to be used in a later effectiveness trial. In addition, the study will determine the feasibility and acceptability of the mobile app.

Recruitment. Participants will be recruited from patient waiting rooms and medical offices of the NMCSD and pharmacy waiting areas using two approaches. The first approach is using flyers about the study opportunity that will be posted in the waiting areas, clinics, and pharmacy. The flyer will instruct potential participants to contact the Principal Investigator (PI) to learn more about the study. The second approach is an in-person approach to tell potential participants about the study opportunity. This will occur by having a research team member onsite in the pharmacy waiting room area handing out flyers and asking potential participants if they would be interested in the study. The research team member can explain more about the study, go over the inclusion criteria, and answer any questions. Similarly, when a clinic staff member or provider sees a clinic patient, he or she will hand them a flyer.

When the potential participant contacts the PI about the study, the PI will verbally confirm if the participant meets the inclusion criteria. The PI will also emphasize that participation is voluntary. If they meet the criteria, the PI will then ask for their non-Department of Defense (DoD) email address to communicate with the participant during the study, and to link their surveys over time. Non-DoD email addresses are less likely to contain a person's full name compared to DoD email addresses. However, in the case that the potential participant is uncomfortable using their current non-DoD (personal) email address, the investigators will provide instructions for setting up a new personal email account on Gmail if they would like to create a new email address for the study to further ensure their anonymity. The PI will send an email to the participant with the: (1) consent form in an attachment for their review; (2) a web link to access the survey website; and (3) instructions for creating a new personal email address for the study with a request to send that to the PI.

The PI or study staff will randomly assign the participant to a study condition, which will indicate which survey link or path, specific to the study condition that they will receive, and then the participant will be sent an email. Each email path will have identical consent documentation; however, this method enables the study team to tailor the follow up messaging more easily. The PI will maintain a list of participant emails and their study group assignment for the purpose of sending survey and intervention reminders.

Informed consent plan. The participant will have received a copy of the consent form in the email from the PI. Also, once the participant accesses the web link (for either survey path-intervention group or control group), the first page they will see will be the consent page. If the participant has any questions, the form encourages the participant to contact the PI and ask questions about the research. If the participant consents to participate, they will indicate this on the web-based consent form by clicking the appropriate box ("I consent" or "I do NOT consent"). If "I do NOT consent" is selected, a screen that thanks them for visiting the site will appear along with the standard instruction to close their browser. The participant must also check a box indicating that they attest that their participation is during off-duty, liberty or leave status to continue to the survey.

Procedures. After the subject consents to participate, the website will also present them with a statement that requires the participant to agree, by checking a box, that their participation will only take place during their off-duty time. (The consent form also clearly instructs participants to complete the survey during their off-duty time.)

The surveys will be web-based and the website will be hosted on a Qualtrics server that uses a high-end firewall system, transport layer security, passwords, and encryption.

Participants will be asked to enter their non-DoD email address as a way to link their surveys over time. Then, they will enter their responses online; their data will automatically be saved to a data file. Measures will be taken to protect the email addresses and survey data collected. After submitting the baseline survey, participants in the intervention group will get instructions for downloading the app. They will be asked to download the app from the app store (e.g., iOS or Google app store), and they will be given a unique key number to access the app once downloaded. The user will also be required to set up a separate self-selected 4-digit PIN and re-enter it each time they open the app, to further enhance security. Neither the participant's phone number nor any identification that can be used to identify the phone or its user will ever be stored in the app developer's server.

While the intervention participants will see the above described download instructions prior to this step, control group participants will be directed to the gift code page immediately after completing their baseline survey. At this gift code page all participants will be presented with instructions on how to get their electronic gift code as a thank-you for their time.

The baseline survey and the 2 follow-up surveys will take about 40 minutes each to complete. The subject will be notified via email about when to complete the baseline, 1-month, and 3-month surveys. There will be an initial request to complete each survey, followed by 2 reminders.

Measures. The data collected for this study will be self-reported survey data collected at baseline, 1 month and 3 months after baseline.

The main outcome measure is the Current Opioid Misuse Measure as an indicator of the risk of opioid misuse. The secondary outcome measures are: the Pain Medication Questionnaire (also an indicator of risk of prescription drug misuse), prescription drug attitudes, knowledge related to prescription drug misuse and preparedness to talk about misuse. All outcomes will be measured as the change from baseline to the follow-up surveys (at 1 and 3 months). These are listed in the Outcomes Measures section of this record; however, additional scale information is described here:

Risk of opioid misuse. The Current Opioid Misuse Measure (COMM) (Butler et al., 2007) was used to measure risk for opioid prescription drug misuse. It measures 17 misuse behaviors over the past 30 days for those currently taking medications.

Risk of misuse. Risk for prescription drug misuse was measured using a 5-item scale that was adapted from a brief scale previously used by Morasco and Dobscha (2008), which is actually a subset of the Pain Medication Questionnaire (PMQ) scale (Adams et al., 2004). The original scale was created to screen for prescription drug misuse among chronic pain patients undergoing opioid therapy, and the shortened scale was created for use among a military veteran population. The present scale includes items such as, "I get pain medication from more than one doctor in order to have enough medication for my pain" and "at times I need to take medication more often than it is prescribed in order to relieve my pain."

Attitudes. Attitudes were assessed in 2 ways. First, the 8-item Prescription Drug Attitudes Questionnaire (PDAQ) (Bodenlos et al., 2014) was adapted by the investigators for the military for this study. Second, the investigators developed 22 prescription drug misuse-related attitude items that specifically aligned with the app's main messages.

Knowledge. Twenty-three multiple choice knowledge items will assess the participant's level of knowledge of the definition of misuse and related educational points.

Preparedness to talk about misuse. Two investigator-developed items were used to assess the level of preparedness to talk to others (i.e., chain of command, doctor) about concerns related to one's own possible prescription drug misuse, In addition, two other investigator-developed items were used to assess the level of preparedness to talk to others about their (e.g., fellow service member, spouse) possible misuse.

Additional measures include: medication use and pain; mental well-being (using the PC-PTSD (Prins et al., 2003) based on the PTSD Checklist (Weathers, Litz, Herman, Huska, & Keane, 1993); PHQ-4 (Kroenke, Spitzer, Williams, & Lowe, 2009); and the Defense and Veterans Brain Injury Center TBI screening tool (Schwab, Baker, Ivins, et al., 2006)); and participant's demographics.

In addition, experimental group participants only will receive 21 items about their experience with the app in the 1-month and 3-month surveys. These items will assess time spent using the app, ease of use, overall satisfaction with the app, usefulness of particular sections, relevance of the content, etc. Also, aggregated data on app page views and navigation patterns will be assessed. This aggregated usage information is collected securely and anonymously for research purposes.

Statistical analysis plan:

Results will be analyzed using a 2 x 3 (group: experimental/control, by time: baseline/1-month/3-month), repeated measures analyses of variance (ANOVA) to examine the potential effectiveness of the program over the 3-month study period. Categorical outcomes will be analyzed using generalized linear mixed models for binary outcomes. Group by time interactions will be examined for any evidence of improvement where greater positive changes in risk for misuse and related outcomes for the experimental group compared to the control group are observed. In addition, descriptive statistics will be used to assess the sample and to examine experimental group participants' satisfaction with and use of the app. Attrition analyses using independent t-tests and Chi-square tests will be carried out among the total sample, as well as by group to examine differences in participant characteristics among attriters and non-attriters. An alpha level of 5% will be assumed in all statistical tests. All analyses will be conducted using IBM SPSS Statistics 19.0.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older (up to 55 years old)
* On active-duty status
* In the Navy or Marine Corps
* Currently prescribed a medication with the potential for misuse
* Owns a smartphone

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne L Hurtado, MPH, Principal Investigator — Naval Health Research Center
Locations (1):
- Naval Health Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams LL, Gatchel RJ, Robinson RC, Polatin P, Gajraj N, Deschner M, Noe C. Development of a self-report screening instrument for assessing potential opioid medication misuse in chronic pain patients. J Pain Symptom Manage. 2004 May;27(5):440-59. doi: 10.1016/j.jpainsymman.2003.10.009. PMID 15120773
- [Background] Butler SF, Budman SH, Fernandez KC, Houle B, Benoit C, Katz N, Jamison RN. Development and validation of the Current Opioid Misuse Measure. Pain. 2007 Jul;130(1-2):144-56. doi: 10.1016/j.pain.2007.01.014. Epub 2007 May 9. PMID 17493754
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Background] Morasco BJ, Dobscha SK. Prescription medication misuse and substance use disorder in VA primary care patients with chronic pain. Gen Hosp Psychiatry. 2008 Mar-Apr;30(2):93-9. doi: 10.1016/j.genhosppsych.2007.12.004. PMID 18291290
- [Background] Prins A, Ouimette P, Kimerling R, Cameron RP, Hugelshofer DS, Shaw-Hegwer J, …Sheikh JI. (2003). The primary care PTSD screen (PC-PTSD): development and operating characteristics. Primary Care Psychiatry, 9(1), 9-14.
- [Background] Bodenlos, J. S., Malordy, A., Noonan, M., Mayrsohn, A., & Mistler, B. (2014). Prescription Drug Attitudes Questionnaire: Development and Validation. Psychology, 5(14), 1687-1693.
- [Background] O'Neill AK. Norms, Attitudes, Perceptions, and Intentions for Benzodiazepine Prescription Drug Abuse among Adolescents (2011). Master's Theses and Doctoral Dissertations. Paper 422.
- [Background] Schwab K, Baker G, Ivins B, Sluss-Tiller M, Lux W, Warden D. (2006). The Brief Traumatic Brain Injury Screen (BTBIS): Investigating the validity of a self report instrument for detecting traumatic brain injury (TBI) in troops returning from deployment in Afghanistan and Iraq. Neurology, 66, A235.
- [Background] Weathers FW, Litz BT, Herman DS, Huska JA, Keane TM. (1993, October). The PTSD Checklist (PCL): Reliability, validity, and diagnostic utility. Paper presented at the annual meeting of the International Society of Traumatic Stress Studies, San Antonio, TX. Retrieved from http://www.pdhealth.mil/library/downloads/pcl_sychometrics.doc.

RESULTS

PARTICIPANT FLOW:
Groups:
- App + Treatment as Usual: The experimental group will be provided with the prescription drug-abuse education smartphone application in addition to treatment as usual. The educational mobile phone app focuses on helping military members reduce their risk for prescription drug misuse.
  As a patient-centered prevention effort, this brief intervention in a mobile phone app format focuses on helping military members reduce their risk for prescription drug misuse. It contains modules to: (1) assess risk for misuse and related behavioral health concerns; (2) provide individualized feedback on risk level; (3) store information on current medications and look up drug interaction and related information; (4) enhance communication and decision-making skills within healthcare and other interpersonal contexts by providing interactive scenarios; (5) teach about the risks of prescription drug misuse; and (6) provide available resources for help with prescription drug misuse.
Period: 1-month to 3-month
Arm/Group | App + Treatment as Usual | Treatment as Usual
Started | 41 | 39
Completed | 35 | 39
Not Completed | 6 | 0
Period: Baseline to 3-month
Arm/Group | App + Treatment as Usual | Treatment as Usual
Started | 35 | 39
Completed | 31 | 39
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- App + Treatment as Usual: The experimental group will be provided with the prescription drug-abuse education smartphone application in addition to treatment as usual. This educational mobile phone app focuses on helping military members reduce their risk for prescription drug misuse.
  As a patient-centered prevention effort, this brief intervention in a mobile phone app format focuses on helping military members reduce their risk for prescription drug misuse. It contains modules to: (1) assess risk for misuse and related behavioral health concerns; (2) provide individualized feedback on risk level; (3) store information on current medications and look up drug interaction and related information; (4) enhance communication and decision-making skills within healthcare and other interpersonal contexts by providing interactive scenarios; (5) teach about the risks of prescription drug misuse; and (6) provide available resources for help with prescription drug misuse.
- Total: Total of all reporting groups
Arm/Group | App + Treatment as Usual | Treatment as Usual | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 39 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 24 | 26 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 14
  Not Hispanic or Latino | 29 | 35 | 64
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 9 | 14
  White | 19 | 21 | 40
  More than one race | 7 | 6 | 13
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 41 | 39 | 80
Branch of Service [Count of Participants; unit: Participants]
  Navy | 31 | 35 | 66
  Marine Corps | 10 | 4 | 14
Education [Count of Participants; unit: Participants]
  less than high school | 1 | 1 | 2
  Finished high school | 4 | 5 | 9
  Finished high school and some college | 36 | 33 | 69
Deployment History [Count of Participants; unit: Participants]
  Ever Deployed | 31 | 24 | 55
  Never Deployed | 10 | 15 | 25

OUTCOME MEASURES:

1. Primary Outcome: Current Opioid Misuse Measure (COMM)
Description: Mean COMM scale score as an indicator of risk for opioid prescription drug misuse. It measures 17 misuse behaviors over the past 30 days for those currently taking medications. Scores can range from 0-4 with higher scores indicating a worse outcome.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App + Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 35 | 39
score on a scale
  Baseline mean | .72 (.37) | .71 (.49)
  1 month mean | .62 (.47) | .63 (.40)
Statistical Analysis 1: Comparison: App + Treatment as Usual vs Treatment as Usual; Test type: Superiority; p = .72, ANOVA — This p-value is the for the group by time (group: intervention/control, by time: baseline/1 month) interaction

2. Secondary Outcome: Pain Medication Questionnaire (PMQ) Shortened Scale
Description: Mean PMQ scale score as an indicator of prescription drug misuse. This 5-item scale was adapted from a brief scale previously used by Morasco and Dobscha (2008), which is actually a subset of the Pain Medication Questionnaire (PMQ) scale (Adams et al., 2004). The original scale was created to screen for prescription drug misuse among chronic pain patients undergoing opioid therapy, and the shortened scale was created for use among a military veteran population. Scale ranges from 1-5 with higher scores indicating a worse outcome.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App + Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 35 | 39
score on a scale
  Baseline PMQ Mean | 1.34 (.48) | 1.43 (.49)
  1 month PMQ Mean | 1.37 (.43) | 1.41 (.49)
Statistical Analysis 1: Comparison: App + Treatment as Usual vs Treatment as Usual; Test type: Superiority; p = .598, ANOVA — This p-value is the for the group by time (group: intervention/control, by time: baseline/1 month) interaction

3. Secondary Outcome: Prescription Drug Misuse-related Attitudes
Description: A scale score for items from the 8-item Prescription Drug Attitudes Questionnaire (PDAQ; Bodenlos et al., 2014), which were adapted by the investigators for the military. The scores range from 1-5 with higher scores indicating a worse outcome.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App + Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 33 | 39
score on a scale
  Baseline PDAQ mean | 1.81 (.58) | 1.82 (.75)
  1 month PDAQ mean | 1.84 (.62) | 1.84 (.75)
Statistical Analysis 1: Comparison: App + Treatment as Usual vs Treatment as Usual; Test type: Superiority; p = .954, ANOVA — This p-value is the for the group by time (group: intervention/control, by time: baseline/1 month) interaction

4. Secondary Outcome: Prescription Drug Misuse-related Knowledge
Description: Mean number of correct knowledge items. Twenty-three multiple choice knowledge items assessed the participant's level of knowledge of the definition of misuse and related educational points. Possible range is 0-23 with higher scores reflecting higher knowledge levels.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: correct items
Arm/Group | App + Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 32 | 39
correct items
  Baseline knoweldge mean | 14.09 (1.84) | 13.26 (2.52)
  1 month knowledge mean | 13.69 (2.05) | 13.44 (2.27)
Statistical Analysis 1: Comparison: App + Treatment as Usual vs Treatment as Usual; Test type: Superiority; p = .167, ANOVA — This p-value is the for the group by time (group: intervention/control, by time: baseline/1 month) interaction

5. Secondary Outcome: Preparedness to Talk About Misuse
Description: Two investigator-developed items were used to assess the level of preparedness to talk to others (i.e., chain of command, doctor) about concerns related to one's own possible prescription drug misuse. The scale ranged from 1-5 with higher scores indicating a better outcome.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App + Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 35 | 39
score on a scale
  Baseline preparedness mean | 3.24 (1.14) | 3.41 (1.12)
  1 month preparedness mean | 3.81 (.97) | 3.36 (1.19)
Statistical Analysis 1: Comparison: App + Treatment as Usual; Test type: Superiority; p = .022, ANOVA — This p-value is the for the group by time (group: intervention/control, by time: baseline/1 month) interaction

ADVERSE EVENTS:
Time Frame: Throughout the duration of participation which would be 4 months for any given participant.
Arm/Group | App + Treatment as Usual | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39

LIMITATIONS AND CAVEATS:
While the sample size was large enough for a pilot of the efficacy of the app based upon calculations, it may have been too limited to determine if there were subgroups of the population for whom the app might have been a more effective intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT03165175/Prot_SAP_ICF_000.pdf